CLINICAL TRIAL: NCT03480347
Title: The BLF Early COPD Development Partnership Grant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: Queen's University, Belfast (Other); University of Southampton (Other); University of Birmingham (Other); University College, London (Other); University of Nottingham (Other); University of Edinburgh (Other); University of Manchester (Other); Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS Project ID: 206796
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples will be collected to determine full Blood count,. Blood serum, plasma and a blood pellet (DNA) will be stored for further analysis of markers of inflammation and infection.
  * Sputum samples (either spontaneous or induced) will be collected and stored and used for microbiome studies, inflammatory markers, and pathogen detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most existing medical research has focused on patients with well-established COPD and poor lung function. Whilst this is important because such patients have lots of symptoms and problems, in some respects a better way of reducing health problems in the future would be to develop a strategy which focuses on patients with milder disease, and identifies which ones will go on to develop more severe problems and why these problems occur. The research in this application is designed to investigate these issues.

The main objective of the Partnership is to study the very early stages of the development of COPD. The investigators will do this by recruiting a novel cohort of smokers (age 30-45), in whom the investigators will follow the trajectories of lung function decline to identify prospectively those at risk of excess decline. This programme forms a unique UK consortium of 8 academic centres with excellent high quality publication records and broad experience in mechanistic, translational, clinical and epidemiological studies in COPD with key capabilities including primary care.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all the following criteria:

* Informed Consent: Subjects must give their signed and dated written informed consent to participate
* Gender: Male or female subjects
* Age: 30-45 years of age at screening
* Smokers of at least 10 pack years
* Have either normal lung function or mild lung function abnormalities
* Subject groups will have one of the following:

  * A. Subjects (smokers) with mild airflow limitation defined as an FEV1/FVC ratio <lower limit of normal and FEV1 > 80% of predicted normal and no symptoms. This group will make up at least 30% of the total cohort.
  * B. Subjects (smokers) with mild airflow limitation as defined above and presence of respiratory symptoms defined as presence of chronic cough and/or chronic sputum and/or breathlessness equivalent to mMRC Grade 1 or higher. This group will make up no more than 25% of the total cohort.
  * C. Subjects (smokers) with normal lung function defined as FEV1/FVC > lower limit of normal and FEV1 > 80% of predicted normal, with or without symptoms. This group will make up at least 30% of the total cohort.

Exclusion Criteria:

* Individuals currently diagnosed and treated for asthma will be excluded from the study, but individuals with a past history of childhood wheezing and of asthma may be included provided that they did not previously receive regular maintenance inhaled therapy with inhaled corticosteroids'
* Subjects with another known chronic respiratory disease - other than mild airflow limitation as defined above, predominantly cannabis or shisha smokers
* Subjects with autoimmune disease, diabetes, hypertension, thyroid disease or bronchiectasis, significant cardio-renal disease (including significant hypertension, atrial fibrillation, Hypertrophic Cardiomyopathy, significant cardiovascular disease), Malignancies.
* Clinically relevant abnormal laboratory values available at the screening assessment that could interfere with the objectives of the study or safety of the volunteer.
* Subjects who are actively enrolled in an interventional clinical trial
* Subjects with BMI >35
* Female participants who are pregnant or breastfeeding.

Ages: 30 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: You can take part in the study if you are 30-45 years of age and you are a current smoker (smokers of at least 10 pack years).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Annual change in lung function | Three years
  assessed by post-bronchodilator at 6 monthly intervals over a 3 year period.
Annual change in lung function | Three years
  assessed by body box plethysmography at 6 monthly intervals over a 3 year period.

SECONDARY OUTCOMES:
Lung tissue attenuation and airway dimensions | Three years
  determined by CT-Scanning
Lung tissue attenuation and airway dimensions | Three years
  Assessed by full blood and differential counts
Lung tissue attenuation and airway dimensions | Three years
  Assessed by prevalence of chronic bronchitis as determined by MRC Bronchitis Questionnaire
Lung tissue attenuation and airway dimensions | Three years
  Assessed by respiratory symptoms, as determined by CAT Questionnaire
Lung tissue attenuation and airway dimensions | Three years
  Assessed by dyspnoea as determined by MRC Dyspnoa Scale
Lung tissue attenuation and airway dimensions | Three years
  Assessed by respiratory infections as determined by Respiratory Infection Questionnaire
Lung tissue attenuation and airway dimensions | Three years
  Assessed by depression and anxiety as determined by Hospital Anxiety Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Ritchie AI, Donaldson GC, Hoffman EA, Allinson JP, Bloom CI, Bolton CE, Choudhury G, Gerard SE, Guo J, Alves-Moreira L, McGarvey L, Sapey E, Stockley RA, Yip KP, Singh D, Wilkinson T, Fageras M, Ostridge K, Jons O, Bucchioni E, Compton CH, Jones P, Mezzi K, Vestbo J, Calverley PMA, Wedzicha JA; British Early COPD Network (BEACON) Cohort Investigators. Structural Predictors of Lung Function Decline in Young Smokers with Normal Spirometry. Am J Respir Crit Care Med. 2024 May 15;209(10):1208-1218. doi: 10.1164/rccm.202307-1203OC. PMID 38175920